CLINICAL TRIAL: NCT02523326
Title: Design of a Protocol for Obtaining Genomic DNA From Saliva Using Mouthwash: Samples Taken From Patients With Periodontal Disease
Brief Title: Design of a Protocol for Obtaining Genomic DNA From Saliva
Acronym: DPOGDNAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Interdisciplinario de Ciencias de la Salud Unidad Santo Tomás (Other)
Responsible Party: Principal Investigator, ÁNGEL CHÁVEZ MENDOZA, PHD STUDENT/professor, Centro Interdisciplinario de Ciencias de la Salud Unidad Santo Tomás
Other Study IDs: CentroICSUT
Record Dates: First submitted 2015-08-04; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Periodontal Disease "Unrecognized Condition"
Keywords: Genomic DNA; chronic periodontitis; saliva; mouthwash; PCR; genotyping; sequencing
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the extraction of high quality genomic DNA from saliva samples obtained with mouthwash.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group A: Each patient was instructed how to prepare for saliva sampling. Patients were instructed to rinse their mouth vigorously with 10 ml of mouthwash during 30 s, then spit it into the tube and the extraction of DNA was performed at distinct times: group A at 10 days
  Interventions: Device: saliva samples obtained with mouthwash
- Group B: Each patient was instructed how to prepare for saliva sampling. Patients were instructed to rinse their mouth vigorously with 10 ml of mouthwash during 30 s, then spit it into the tube and the extraction of DNA was performed at distinct times: group B at 20 days
  Interventions: Device: saliva samples obtained with mouthwash
- Group C: Each patient was instructed how to prepare for saliva sampling. Patients were instructed to rinse their mouth vigorously with 10 ml of mouthwash during 30 s, then spit it into the tube and the extraction of DNA was performed at distinct times: group C at 30 days
  Interventions: Device: saliva samples obtained with mouthwash

INTERVENTIONS:
Device: saliva samples obtained with mouthwash — saliva samples obtained with mouthwash

SUMMARY:
Objective The aim of this study was to test a protocol for the extraction of high quality genomic DNA from saliva samples obtained with mouthwash and taken from patients with periodontal disease.

Materials and methods Saliva samples were taken from 60 patients, then stored at room temperature. DNA extraction was carried out at distinct post-sampling times (10, 20 and 30 days). Evaluation of genomic DNA was performed with spectrophotometry, electrophoresis, and PCR genotyping and sequencing.

DETAILED DESCRIPTION:
Materials and methods 2.1. Patients The study was conducted with 60 patients diagnosed with severe chronic periodontitis in the Periodontic Clinic of the Interdisciplinary Health Sciences Center (Santo Tomás Unit), National Polytechnic Institute. The protocol of this study was approved by the Research and Bioethics Committee of the School of Medicine. National Polytechnic Institute. Informed consent was obtained from all participants included in the study, who signed the appropriate form allowing for the collection of saliva samples and the extraction of genomic DNA. Ethical norms for research on human beings, established by the Declaration of Helsinki (1975; updated most recently in 2008) were strictly followed. Each patient was instructed how to prepare for saliva sampling, which involved brushing their teeth at least 2 h previously and abstaining from eating or drinking anything.

2.2. Taking the sample In a tube of 50 ml were placed 10 ml mouthwash (Listerine Cool Mint, Johnson & Johnson, 21.6% alcohol). Patients were instructed to rinse their mouth vigorously with this quantity of mouthwash during 30 s, then spit it into the tube. Once collected, the samples were stored at room temperature (20°C - 24°C). The 60 samples were divided into 3 groups (n=20), and the extraction of DNA was performed at distinct times: group A at 10 days, group B at 20 days and group C at 30 days.

2.3. DNA extraction To separate the mouthwash, the tube was centrifuged during 10 min at 10750x g. The supernatant was poured out and the cellular pellet washed with 1 ml of PBS, resuspended in the vortex for 30 s, and transferred to a new 2 ml tube. It was then centrifuged for 5 min at 2000x g, the supernatant poured out, and the pellet washed with 1.5 ml of PBS and resuspended in the vortex for 30 s. To this solution was added a 1 ml solution of lysis of nucleated cells (Wizard® Genomic DNA Purification Kit) before being shaken for 20 s, followed by incubation at 37 °C for 10 min. After adding 300 µl of protein precipitator solution (Wizard® Genomic DNA Purification Kit), the mixture was placed on ice for 5 min and then centrifuged at 15000x g for 3 min. The supernatant was put in a 1.5 ml tube containing 600 µL cold Isopropanol and homogenized gently, then centrifuged at 15000x for 3 min. The supernatant was poured out and 600 µL of 70% ethanol were added to a fresh preparation, which was centrifuged at 15000x g for 3 min. The supernatant was poured out and the tube was completely dried at room temperature. Finally, 100 µL rehydration solution (Wizard® Genomic DNA Purification Kit) was added and the mixture was incubated at 64 °C for 1 h before storing the samples at -20 °C to await further processing.

2.4. DNA evaluation Evaluation of the concentration and purity of DNA was determined by spectrophotometry with an ACT-GENE ASP-3700 spectrometer. The concentration of DNA was evaluated at 260 nm, while purity was estimated with the ratios of 260/203 and 260/280. The integrity of genomic DNA was assessed in a 0.8% agarose gel in 1% TBE (89 mM Tris Borate, 89 mM boric acid, 2 mM EDTA) by electrophoresis, and then the DNA was visualized with Gel-Red and read under UV light. DNA extracted from blood samples was used as the positive control.

2.5. PCR The PCR reaction was carried out in an Eppendorf Mastercycler® Personal apparatus with the HotStarTaq ® Master Mix Qiagen kit (No. de Cat 203445), following the manufacturer's instructions. To verify the quality and species (human) of the DNA extracted, primers were designed for the rs679620 polymorphism (forward 5´- ggg gCT TAA ggC ACA TgA gT-3; reverse 5´- ACT TCg ggA TgC CAg gAA Ag - 3´; Tm: 56°C, 40 cycles) that amplified a product of 485 bp. The final PCR product was evaluated with a 2% agarose gel. DNA extracted from blood samples was used as a positive control.

2.6. Sequencing To further verify the quality and species of the DNA obtained, the product resulting from PCR was sequenced with an Applied Biosystems 3130 sequencer and the BigDye® Terminator v3.1 Cycle Sequencing kit, following the manufacturer's instructions. Data were analyzed with Geneious version 7.1.3 software [23], using the NC_000011.10 sequence as the reference.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with severe chronic periodontitis
* who signed the appropriate form allowing for the collection of saliva samples and the extraction of genomic DNA

Exclusion Criteria:

* NO diagnosed with severe chronic periodontitis
* NO signed the appropriate form allowing for the collection of saliva samples and the extraction of genomic DNA

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients diagnosed with severe chronic periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
DNA | 10 days [group A], 20 days [group B], 30 days [group C]
  high quality genomic DNA from saliva samples obtained with mouthwash.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Buentello Volante, Doctorate, Principal Investigator — Instituto de Oftalmología "Conde de Valenciana".; María Esther Ocharán Hernández, Doctorate, Principal Investigator — Escuela Superior de Medicina, Instituto Politécnico Nacional; Claudia Camelia Claudia Camelia Calzada Mendoza, Doctorate, Principal Investigator — Escuela Superior de Medicina, Instituto Politécnico Nacional; Arturo Flores Pliego, Doctorate, Principal Investigator — Instituto Nacional de Perinatología; Héctor A. Baptista Gonzalez, Doctorate, Principal Investigator — Instituto Nacional de Perinatología; Higinio Estrada Juárez, Doctorate, Study Director — Instituto Nacional de Perinatología
Locations (1):
- Angel Chavez Mendoza, México, D.f., Mexico